CLINICAL TRIAL: NCT07214350
Title: Sex Differences in Barriers and Participation in Physical Activity During and Following Cardiac Rehabilitation
Acronym: SPARC
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00118596; 1K01HL177266-01A1 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Rehabilitation; Heart Disease
Keywords: Physical Activity; Sex Differences
MeSH Terms: conditions — Heart Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults participating in cardiac rehabilitation: Physical activity and functional fitness will be measured during cardiac rehabilitation, right after completion of cardiac rehabilitation, and 6 months later.

SUMMARY:
The SPARC study will measure physical activity and functional fitness during cardiac rehabilitation, right after completion of cardiac rehabilitation, and 6 months later. This will help investigators learn if men and women maintain physical activity levels and functional fitness differently during and after they complete cardiac rehabilitation. Participants in this study will have three in-person study visits and may complete two qualitative interviews over a 10-month study period. The greatest risks during the study include physical discomfort, falling, and/or shortness of breath during the fitness testing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Enrolled in cardiac rehabilitation within the last month
* Own a smartphone or tablet for mobile application download

Exclusion Criteria:

* Planned relocation during the study period out of the local area
* Planned medical procedure within the study period that may limit physical activity (i.e., joint replacement)
* End-stage kidney disease
* Impairment from stroke, injury, or other medical conditions that would prevent participation in or completion of the protocol
* Heart transplant
* Use of a left ventricular assist device
* Pregnant or intending to become pregnant during the study period
* Any other illness that, in the opinion of the study physician, would negatively impact or mitigate participation in or completion of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults participating in cardiac rehabilitation
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Average Daily Step Count | Baseline, 3 months, 9 months
  Calculated as an average of daily steps achieved over the previous week at each timepoint.

SECONDARY OUTCOMES:
Average moderate-to-vigorous physical activity minutes per week | 9 months
  Self-reported moderate-to-vigorous-intensity physical activity minutes per week using the Paffenbarger Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A. Collins-Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will produce demographic, clinical and psychological obtained at baseline, 3-, and 9 months following participant enrollment. Data will be collected from a maximum of 186 research participants (total enrollment goal n = 150). To protect research participant identities, data will be de-identified; only de-identified data will be made available for sharing. Data collection will be performed at the Center for Living Campus - part of the Duke Molecular Physiology Institute - at the Duke University School of Medicine. In this proposed project for data relevant to the Specific Aims, the cleaned, item-level spreadsheet data will be shared openly, along with example transformations from initial raw data. Final files used to generate specific analyses to answer the Specific Aims and related results will also be shared. The rationale for sharing only cleaned data is to foster ease of data reuse.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared either at the time of publication or at the end of the performance period, whichever comes first.
Access Criteria: The Duke Library DRD provides searchable study-level metadata for dataset discovery, assigns DOIs as persistent identifiers, and has a robust preservation plan to ensure long-term access. Data will be discoverable online through a standard web search of the study-level metadata as well as the persistent pointer from the DOI to the dataset. The RDR will assign appropriate metadata (Dublin Core) for discoverability and provide a DataCite Digital Object Identifier (DOI) for persistent access and unique identification of the data, all data in the RDR are findable with standard indexing tools and included in Google Datasets and DataCite Commons.